CLINICAL TRIAL: NCT01736358
Title: Evaluating Post-operative Pain Management Efficacy of Intra Nasal Ketorolac in Ambulatory Urological Surgeries-A Randomized Double-blinded Placebo Controlled Study
Brief Title: The Use of Intranasal Ketoralac for Pain Management (Sprix)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed futility of primary endpoint
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Singh Nair, Associate Professor, Dept of Urology, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 12-02-244
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain Management; Urolithiasis
Keywords: Sprix; Intranasal ketoralac; Ketoralac; Urolithiasis; Kidney stone; Uretal stone; Ureteroscopic removal of stones; URS; Pain management; Pain
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Agnosia; Pain | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Ketoralac (Experimental): A single dose of Sprix (31.5 mg) will be administered to patients 20 minutes before the end of surgery. 15.75 mg of Sprix will be sprayed in each nostril.
  Interventions: Drug: Intranasal Ketoralac
- Placebo (Placebo Comparator): A single dose of placebo will be administered 20 minutes before the end of surgery. 15.75 mg of the placebo will be sprayed in each nostril.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Ketoralac — 15.75 mg of Sprix in each nostril 20 minutes before end of surgery
  Other Names: Sprix
  Arms: Intranasal Ketoralac
Drug: Placebo — 15.75 mg of placebo will be administered in each nostril 20 minutes before the end of surgery
  Arms: Placebo

SUMMARY:
Despite an overall reduction in the perioperative complication rate, post operative pain management after ureteroscopic removal of stones (URS) remains a major factor delaying discharge of patients. The investigators hypothesize that perioperative usage of intranasal ketorolac will provide a reduction in post operative opioid requirements, better post operative pain control, higher anesthesia satisfaction and faster recovery.

DETAILED DESCRIPTION:
The prevalence and incidence of urolithiasis, or kidney stone disease, are increasing in the general population. Life-time incidence of urolithiasis is estimated to be between 5%- 12%. The treatment of kidney stones depends on stone type and size, symptom severity, and the presence of obstruction.

URS is a common ambulatory procedure as improved technological advances and increased clinical utilization have helped decrease postoperative complications. Despite an overall reduction in the perioperative complication rate, post operative pain management after URS remains a major factor delaying discharge of patients.

Post operative pain after URS is usually treated with opioids and non steroidal anti inflammatory drugs. Intranasal ketorolac (SprixTM) is an FDA approved pain formulation for short term management (5 days) of moderate to moderately severe pain that requires analgesia at the opioid level. The efficacy of intranasal ketorolac formulation was demonstrated in placebo-controlled studies in patients following major surgeries.

The primary objective of the study is to evaluate the role perioperative usage of single-dose of intranasal ketorolac on immediate post operative opioid requirements. Secondary objectives of the study are to (a) evaluate the post operative pain score 30 minutes after surgery, 1 hour after surgery, and 2 hours after surgery, (b) find the incidence of immediate (until discharge) and 24hrs post operative side effects in the target population, (c) find the level of anesthesia satisfaction in the target population, (d) find the time to discharge in the target population, (e) compare the two groups post anesthesia discharge score.

ELIGIBILITY:
Inclusion Criteria:

* Ureteroscopic stone removal surgeries with stenting
* Age ≥ 18 years and < 65 years
* Stable patient with stable vital signs
* Mentally competent and is able to understand consent form

Exclusion Criteria:

* Unstable patients
* Patients with multiple trauma sites
* Patients with allergies to ketorolac or any of the components in the nasal spray preparation
* Patients with active peptic ulcer disease
* History of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs
* Renal disease or at risk for renal failure due to volume depletion
* Pregnant or nursing mothers
* Nasal abnormality or illness that could affect the absorption of intranasal medication (such as: nasal discharge, rhinitis, acute upper respiratory infection, acute epistaxis, nasal polyp, nasal tumor)
* Any other contraindication to the use of Sprix, or in whom use of Sprix would not be consistent with the approved package insert

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Singh Nair, MD, Study Director — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center- Weiler Division, The Bronx, New York, United States

REFERENCES:
- [Background] Saigal CS, Joyce G, Timilsina AR; Urologic Diseases in America Project. Direct and indirect costs of nephrolithiasis in an employed population: opportunity for disease management? Kidney Int. 2005 Oct;68(4):1808-14. doi: 10.1111/j.1523-1755.2005.00599.x. PMID 16164658
- [Background] Pak CY, Resnick MI, Preminger GM. Ethnic and geographic diversity of stone disease. Urology. 1997 Oct;50(4):504-7. doi: 10.1016/s0090-4295(97)00307-5. PMID 9338722
- [Background] Peschel R, Janetschek G, Bartsch G. Extracorporeal shock wave lithotripsy versus ureteroscopy for distal ureteral calculi: a prospective randomized study. J Urol. 1999 Dec;162(6):1909-12. doi: 10.1016/S0022-5347(05)68066-4. PMID 10569535
- [Background] Tiselius HG. Epidemiology and medical management of stone disease. BJU Int. 2003 May;91(8):758-67. doi: 10.1046/j.1464-410x.2003.04208.x. PMID 12709088
- [Background] Erhard M, Salwen J, Bagley DH. Ureteroscopic removal of mid and proximal ureteral calculi. J Urol. 1996 Jan;155(1):38-42. PMID 7490892
- [Background] Cheung MC, Lee F, Leung YL, Wong BB, Chu SM, Tam PC. Outpatient ureteroscopy: predictive factors for postoperative events. Urology. 2001 Dec;58(6):914-8. doi: 10.1016/s0090-4295(01)01445-5. PMID 11744457
- [Background] Bromwich EJ, Lockyer R, Keoghane SR. Day-case rigid and flexible ureteroscopy. Ann R Coll Surg Engl. 2007 Jul;89(5):526-8. doi: 10.1308/003588407X187676. PMID 17688729
- [Background] Ahn ST, Kim JH, Park JY, Moon du G, Bae JH. Acute postoperative pain after ureteroscopic removal of stone: incidence and risk factors. Korean J Urol. 2012 Jan;53(1):34-9. doi: 10.4111/kju.2012.53.1.34. Epub 2012 Jan 25. PMID 22323972
- [Background] Moodie JE, Brown CR, Bisley EJ, Weber HU, Bynum L. The safety and analgesic efficacy of intranasal ketorolac in patients with postoperative pain. Anesth Analg. 2008 Dec;107(6):2025-31. doi: 10.1213/ane.0b013e318188b736. PMID 19020154
- [Background] McAleer SD, Majid O, Venables E, Polack T, Sheikh MS. Pharmacokinetics and safety of ketorolac following single intranasal and intramuscular administration in healthy volunteers. J Clin Pharmacol. 2007 Jan;47(1):13-8. doi: 10.1177/0091270006294597. PMID 17192497
- [Background] Brown C, Moodie J, Bisley E, Bynum L. Intranasal ketorolac for postoperative pain: a phase 3, double-blind, randomized study. Pain Med. 2009 Sep;10(6):1106-14. doi: 10.1111/j.1526-4637.2009.00647.x. Epub 2009 Jul 6. PMID 19594851
- [Background] Singla N, Singla S, Minkowitz HS, Moodie J, Brown C. Intranasal ketorolac for acute postoperative pain. Curr Med Res Opin. 2010 Aug;26(8):1915-23. doi: 10.1185/03007995.2010.495564. PMID 20557145
- [Background] Grant GM, Mehlisch DR. Intranasal ketorolac for pain secondary to third molar impaction surgery: a randomized, double-blind, placebo-controlled trial. J Oral Maxillofac Surg. 2010 May;68(5):1025-31. doi: 10.1016/j.joms.2009.10.023. Epub 2010 Mar 5. PMID 20207062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intranasal Ketoralac | Placebo
Started | 25 | 25
Completed | 20 | 23
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Ketoralac | Placebo | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 23 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 47 (12.4) | 49 (9.3) | 48 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 10 | 12 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Opioid Requirements
Description: this study will assess the effect of perioperative usage of single-dose of intranasal ketorolac on post operative opioid requirements within 3 hours after surgery.
Time Frame: 3 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Intranasal Ketoralac | Placebo
Number analyzed (Participants) | 20 | 23
mg | 27.43 [23.87 to 51.30] | 30 [22.05 to 48]

2. Secondary Outcome: Post Operative Pain Score
Description: To evaluate the post operative pain score using the Visual Analog Scale (VAS) 30 minutes after surgery. The scale for VAS is 0 is no pain to 10 being the worst pain.
Time Frame: 30 minutes after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intranasal Ketoralac | Placebo
Number analyzed (Participants) | 20 | 23
score on a scale | 4 [0 to 6] | 3.5 [0 to 7.75]

3. Secondary Outcome: Post Operative Pain Score
Description: To evaluate the post operative pain score using the Visual Analog Scale (VAS) 1 hour after surgery. The scale for VAS is 0 is no pain to 10 being the worst pain.
Time Frame: 1 hour after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intranasal Ketoralac | Placebo
Number analyzed (Participants) | 20 | 23
score on a scale | 3.5 [0 to 5.7] | 4.5 [2 to 6.7]

4. Secondary Outcome: Post Operative Pain Scale
Description: To evaluate the post operative pain score using the Visual Analog Scale (VAS) 2 hours after surgery. The scale for VAS is 0 is no pain to 10 being the worst pain.
Time Frame: 2 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intranasal Ketoralac | Placebo
Number analyzed (Participants) | 20 | 23
score on a scale | 4 [0 to 7.7] | 3 [0 to 5]

5. Other Pre Specified Outcome: Incidence of Postoperative Side Effects
Description: To find the incidence of immediate (until discharge) and 24hrs post operative side effects in the target population.
Time Frame: 24 hours after procedure
Measure: Number; unit: number of events
Arm/Group | Intranasal Ketoralac | Placebo
Number analyzed (Participants) | 20 | 23
number of events | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intranasal Ketoralac | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 0/20 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No